CLINICAL TRIAL: NCT05692349
Title: Role of Magnetic Resonance Imaging and Ultrasonography in Evaluation of Muscle Diseases
Brief Title: Magnetic Resonance Imaging and Ultrasonography in Evaluation of Muscle Diseases
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Tayseer Mohamed Hashem Hamza, Resident doctor at assiut university, Assiut University
Other Study IDs: MRI and US in Muscle Disease
Record Dates: First submitted 2022-07-22; First posted 2023-01-20 (Actual); Last update posted 2023-01-20 (Actual); Status verified 2023-01

CONDITIONS: Congenital Myopathy; Acquired Myopathy; Myositis
Keywords: Muscle disease
MeSH Terms: conditions — Myotonia Congenita; Myositis; Muscular Diseases | interventions — Electromyography

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: MRI — MRI will be employed to assess muscle composition, evidence of degeneration or replacement by fat
  Other Names: Muscle Ultrasound; Muscle Biopsy; Neurophysiology (nerve conduction and EMG)

SUMMARY:
This study aims to determine the association between the pathological changes detected by ultrasound and those detected in MRI in muscle diseases of different etiologies.

DETAILED DESCRIPTION:
Enrolled patients will be subjected to the following:

Neuro-imaging Studies:

1. Skeletal Muscle ultrasound:

   The muscle group(s) to be assessed will be determined based on the category of the muscle disease for which the patient is being evaluated. A linear probe of 5-12 megahertz will be used.
2. MRI of the suspected (affected) muscle group by ultrasound. Image acquisition: Selective regional MRI imaging will be done based on the results of muscle ultrasound MRI cuts included are the axial section of conventional T1- and T2-weighted sequences, for the evaluation of muscles' signal intensity and bulk.

Patients will be subjected to both imaging studies to compare their accuracy.

Neurophysiological Studies:

1. Nerve conduction study
2. Electromyogram The interpretation of the neurophysiological studies will be performed by a neuropsychiatry specialist, Department of Neurology, Assiut University Hospital.

ELIGIBILITY:
Inclusion Criteria:

1. A clinical diagnosis of muscle diseases; irrespective of different etiologies
2. Age > 3 years

Exclusion Criteria:

1. Patients with altered muscle anatomy due to severe trauma, tumor or surgery.
2. Severe deformity preventing examination.
3. Age < 3years.
4. Patients with contraindications to MRI as patients with pacemaker, aneurysmal clipping, retained metallic

Min Age: 4 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Muscle Disease of different aetiologies
Sampling Method: Non-Probability Sample
Enrollment: 36 (Estimated)
Dates: Start 2023-01 (Estimated); Primary Completion 2023-09 (Estimated); Study Completion 2024-01 (Estimated)

PRIMARY OUTCOMES:
Percentage of abnormal ultrasound and Magnetic resonance studies separately | through study completion, an average of 1 year
  Abnormal Magnetic resonance study: muscle fat replacement (qualitatively through T1 weighted images, and qualitatively through Mercuric visual grading system), edema ( T2 relaxation time mapping), fibrosis ( magnetic resonance elastography) Abnormal muscle ultrasound study (replacement of healthy muscle with fat and fibrosis, manifested by an increase in echogenicity, visual method based on evaluating echogenicity in relation to other structures and semi-quantitatively)
Association between the results of Skeletal muscle ultrasound (normal vs. abnormal) and the results of MRI (normal vs. abnormal study) | within 6 months after recruitment ends (Recruitment completion is anticipated In Sep 2023)
Association between the individual abnormalities detected by skeletal muscle ultrasound and those detected by MRI. | within 6 months after recruitment ends (Recruitment completion is anticipated In Sep 2023)
Diagnostic accuracy of each modality in reference to the clinical and neurophysiological diagnosis and muscle biopsy. | within 6 months after recruitment ends (Recruitment completion is anticipated In Sep 2023)

CONTACTS AND LOCATIONS:
Overall Officials: Eman A. E. Ahmed, Professor, Study Chair — Assiut University; Sara M. Ahmed, MD, Study Director — Assiut University

REFERENCES:
- [Background] Dahlqvist JR, Widholm P, Leinhard OD, Vissing J. MRI in Neuromuscular Diseases: An Emerging Diagnostic Tool and Biomarker for Prognosis and Efficacy. Ann Neurol. 2020 Oct;88(4):669-681. doi: 10.1002/ana.25804. Epub 2020 Jul 1. PMID 32495452
- [Background] Paoletti M, Pichiecchio A, Cotti Piccinelli S, Tasca G, Berardinelli AL, Padovani A, Filosto M. Advances in Quantitative Imaging of Genetic and Acquired Myopathies: Clinical Applications and Perspectives. Front Neurol. 2019 Feb 11;10:78. doi: 10.3389/fneur.2019.00078. eCollection 2019. PMID 30804884
- [Background] Bugiardini E, Morrow JM, Shah S, Wood CL, Lynch DS, Pitmann AM, Reilly MM, Houlden H, Matthews E, Parton M, Hanna MG, Straub V, Yousry TA. The Diagnostic Value of MRI Pattern Recognition in Distal Myopathies. Front Neurol. 2018 Jun 26;9:456. doi: 10.3389/fneur.2018.00456. eCollection 2018. PMID 29997562
- [Background] Smitaman E, Flores DV, Mejia Gomez C, Pathria MN. MR Imaging of Atraumatic Muscle Disorders. Radiographics. 2018 Mar-Apr;38(2):500-522. doi: 10.1148/rg.2017170112. Epub 2018 Feb 16. PMID 29451848
- [Background] Heckmatt JZ, Dubowitz V, Leeman S. Detection of pathological change in dystrophic muscle with B-scan ultrasound imaging. Lancet. 1980 Jun 28;1(8183):1389-90. doi: 10.1016/s0140-6736(80)92656-2. PMID 6104175
- [Background] Wijntjes J, van Alfen N. Muscle ultrasound: Present state and future opportunities. Muscle Nerve. 2021 Apr;63(4):455-466. doi: 10.1002/mus.27081. Epub 2020 Oct 13. PMID 33051891
- [Background] Albayda J, van Alfen N. Diagnostic Value of Muscle Ultrasound for Myopathies and Myositis. Curr Rheumatol Rep. 2020 Sep 28;22(11):82. doi: 10.1007/s11926-020-00947-y. PMID 32989482
- [Background] Habers GE, Van Brussel M, Bhansing KJ, Hoppenreijs EP, Janssen AJ, Van Royen-Kerkhof A, Pillen S. Quantitative muscle ultrasonography in the follow-up of juvenile dermatomyositis. Muscle Nerve. 2015 Oct;52(4):540-6. doi: 10.1002/mus.24564. Epub 2015 Mar 14. PMID 25557638
- [Background] Pillen S, Morava E, Van Keimpema M, Ter Laak HJ, De Vries MC, Rodenburg RJ, Zwarts MJ. Skeletal muscle ultrasonography in children with a dysfunction in the oxidative phosphorylation system. Neuropediatrics. 2006 Jun;37(3):142-7. doi: 10.1055/s-2006-924512. PMID 16967365